CLINICAL TRIAL: NCT05962619
Title: Arthrocentesis Alone Versus Arthrocentesis With Hyaluronic Acid Injection in Management of Temporomandibular Joint Dysfunction in the Form of Anterior Disc Displacement With Reduction : a Randomized Controlled Trial
Brief Title: Arthrocentesis Alone Versus Arthrocentesis With Hyaluronic Acid Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Hussein Ali, Principle investigator, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AHAI
Record Dates: First submitted 2023-06-12; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Arthrocenteses; Hyaluronic Acid
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome | interventions — Arthrocentesis; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthrocentesis alone (Experimental): Arthrocentesis alone in management of temporomandibular joint dysfunction in the form of anterior disc displacement with reduction.by lavage by normal saline and during the lavage the mandible is moved through opening, excursive, and protrusive movements to facilitate lysis of adhesions.
  Interventions: Procedure: arthrocentesis alone
- arthrocentesis with hyaluronic acid injection (Experimental): arthrocentesis with hyaluronic acid injection in management of temporomandibular joint dysfunction in the form of anterior disc displacement with reduction. after arthrocentesis is completed, lavage is done by hyaluronic acid injection
  Interventions: Procedure: arthrocentesis with hyaluronic acid injection

INTERVENTIONS:
Procedure: arthrocentesis alone — The procedure is done under general anesthesia. The patient is seated inclined at a 45 degree angle with the head turned to contralateral side. The points of needle insertion on the skin, are as follow: a line is drawn from the middle of the tragus to the outer canthus of the eye. The posterior entrance point is located along the canthotragal line, 10 mm from the middle of the tragus line and 2 mm below, the anterior entrance point is placed 10 mm further forward along the line and 10 mm below it . A needle connected to a 10 ml syringe with the Ringer's lactate solution is then inserted into the superior compartment (posterior point), and solution is injected . Another needle is then inserted into the area of articular eminence to enable the free flow of solution through the superior compartment. During the lavage, the mandible is moved through opening, excursive, and protrusive movements to facilitate lysis of adhesions
  Arms: Arthrocentesis alone
Procedure: arthrocentesis with hyaluronic acid injection — in this group Once arthrocentesis is completed, an ampule of sodium HA (Hyalgan 1 ml) is connected to the needle in situ And 0.5 ml injected into the superior joint space. Pressure dressing is placed in site of injection. so We use arthrocentesis hyaluronic acid injection in management of temporomandibular joint dysfunction in the form of anterior disc displacement with reduction
  Arms: arthrocentesis with hyaluronic acid injection

SUMMARY:
Comparison between Arthrocentesis alone arthrocentesis with hyaluronic acid injection in management of temporomandibular joint dysfunction in the form of anterior disc displacement with reduction.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) anterior disc displacement (ADD) is one of the most common TMJ disorders.It can occur in all age groups, with a high prevalence in adolescents .

ADD often presents with clicking, joint pain, a limited range of mouth opening. Furthermore,ADD might lead to osteoarthrosis .

Since ADD of the TMJ can lead to various harmful outcomes, how to manage ADD is considered a key problem for most TMJ experts. It has been difficult for most clinicians to select a suitable method for ADD patients with different grades of severitis ). Initially, these conditions can be managed conservatively by employing techniques such as occlusal splint therapy, physiotherapy, pharmacotherapy and occlusal treatments. If Medical treatment fails, minimally invasive (sodium hyaluronate or corticosteroid infiltrations and arthrocentesis) and invasive treatments (arthroscopy, arthroplasty, arthrotomy, discectomy, condylotomy) are formed ). Sodium hyaluronate is a buffered solution of hyaluronate acid sodium salt, which is an essential component of the cartilage.It acts against the disintegration of the extracellular matrix.It reduces friction, and it features an anti-inflamatory effect. It is indicated for the treatment of osteoarthritic symptoms and inflammatory degenerative joint disease). Intra-articular hyaluronic acid injection provides long-term palliative effects on symptoms and signs of TMJ pain .

ELIGIBILITY:
Inclusion Criteria:

* Adults with age between( 18-45) years
* Both genders
* The cases ciinically have either of ( limitation of mouth opening , pre-auricular pain , headache, temporal, and occipital tenderness ) and radiologically (MRI) diagnosed as ADD with reduction
* The patients have symptom durations for more than 3 months with medical treatment.
* Patients whom did not respond to medical treatment

Exclusion Criteria:

* Previous TMJ surgery or previous arthrocentesis.
* Patients with arthritis or history of condylar trauma
* Patients with degenerative change of the condylar head and with facial asymmetry, retrognathism, or prognathism
* Severe co-morbid conditions (uncontrolled diabetes, Hypertenion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-02 (Estimated)

PRIMARY OUTCOMES:
Mouth opening | Three months
  Maximum inter-incisal opening (MIO): measured by Vernier caliper in millimeters (mm) as the vertical distance between the incisal edges of maxillary and mandibular central incisors. Preoperative and postoperative measurement of MIO would help in evaluation of improvement in mouth opening after arthrocentesis
Tempero mandibular joint pain | One month
  Pain was assessed using visual analogue scale (VAS):
  which ranges from zero to 10 (where zero refers to no pain, 1:3 mild pain, 4:6 moderate pain, 7:9 severe pain and 10 maximum pain) assessing pre and post operative will provide good evidence about effect of arthrocentesis in decrease Tempero mandibular joint pain

SECONDARY OUTCOMES:
Clicking | Three months
  Clicking was assessed as its presence or absence where zero refers to absence of clicking, 1 indicates decrease in sound and frequency of clicking, and 2 indicates presence of clicking.Assessment of clicking showed that there was statistically significant difference between the two groups along the evaluation intervals. There was statistically significant difference between clicking scores at the baseline when compared to the follow-up intervals within both groups

IPD SHARING:
Plan to Share IPD: No